CLINICAL TRIAL: NCT05674006
Title: Ultrasound Guided Sacral Erector Spina Plane Block as a Main Anesthetic Method: Single Center Experience
Brief Title: Ultrasound Guided Sacral Erector Spina Plane Block as a Main Anesthetic Method
Acronym: ESP
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: SamsunU_sakral_ESP
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Anesthesia, Local
Keywords: Anesthesia; ESP; Sacral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this retrospective observational study is to demonstrate investigators' experience of Ultrasound guided Sacral Erector Spina Plane Block as an anesthetic technique in patients underwent sacral plastic and reconstructive surgeries.

The main question[s] it aims to answer are:

* block indication, level
* results, side effects and complications

DETAILED DESCRIPTION:
Erector Spina Plane Block is an interfascial plane block that is performed by injecting the local anesthetic solution between transverse process of the vertebra and erector spina muscle. It is found to be an inexpensive,easily applied, effective and safe technique for chronic pain.(1) Ultrasound guided Erector Spina Plane Block(ESP) is getting more and more widely used for analgesia and as an anesthetic technique.(2,3) Regional anesthesia techniques provide safer, more stable and advantageous anesthetic management, especially in high-risk patients. Ultrasound guided Sacral ESP is described by Tulgar et all.in 2019 and can be used either for analgesia or as an anesthetic technique. (4) In this retrospective study investigators planed to demonstrate one year of experience of this block for sacral plastic and reconstructive surgery. Demographic data of patients who underwent sacral surgery with sacral ESP block, indication of block, level of block, drug dose concentration, effect, side effect and results that were recorded will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* being going for a sacral surgery
* American Society of Anesthesiology status (ASA) 1 - 4

Exclusion Criteria:

* emergency
* ASA-5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ASA1-4 patients of age older than18 going for a sacral surgery
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Block success | up to 1 year
  Effectiveness of Sacral Erector Spinae Plane Block as an Anesthetic technique

SECONDARY OUTCOMES:
Number and amount of required perioperative analgesic/anesthetic drugs | up to 2 hours
  The number and amount of drugs administered will be determined from the anesthesia file records when the patient feels pain or shows dissatisfaction with anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Tulgar, Study Chair — Samsun University
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Unal Artik HA, Gulpinar TO, Halis A, Celebi N. Erector spinae plane block in chronic pain: a retrospective study. Turk J Med Sci. 2022 Aug;52(4):1408-1410. doi: 10.55730/1300-0144.5449. Epub 2022 Aug 10. PMID 36326408
- [Background] Kaya C, Dost B, Tulgar S. Sacral Erector Spinae Plane Block Provides Surgical Anesthesia in Ambulatory Anorectal Surgery: Two Case Reports. Cureus. 2021 Jan 9;13(1):e12598. doi: 10.7759/cureus.12598. PMID 33585088
- [Background] Ahiskalioglu A, Tulgar S, Celik M, Ozer Z, Alici HA, Aydin ME. Lumbar Erector Spinae Plane Block as a Main Anesthetic Method for Hip Surgery in High Risk Elderly Patients: Initial Experience with a Magnetic Resonance Imaging. Eurasian J Med. 2020 Feb;52(1):16-20. doi: 10.5152/eurasianjmed.2020.19224. PMID 32158307
- [Background] Tulgar S, Senturk O, Thomas DT, Deveci U, Ozer Z. A new technique for sensory blockage of posterior branches of sacral nerves: Ultrasound guided sacral erector spinae plane block. J Clin Anesth. 2019 Nov;57:129-130. doi: 10.1016/j.jclinane.2019.04.014. Epub 2019 Apr 15. No abstract available. PMID 30999197